CLINICAL TRIAL: NCT00096733
Title: Adult-to-Adult Living Donor Liver Transplantation Cohort Study
Brief Title: Adult-to-Adult Living Donor Liver Transplantation Study
Acronym: A2ALL-1
Status: Completed | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: American Society of Transplant Surgeons (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: A2ALL; U01DK062498-01 (NIH)
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Cirrhosis; Hepatitis C; Hepatocellular Carcinoma
Keywords: Living donors; Organ procurement; Liver transplantation; Hepatitis C; Hepatocellular carcinoma; Hepatectomy; Liver regeneration; Graft rejection; Quality of life; Informed consent
MeSH Terms: conditions — Fibrosis; Hepatitis C; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood, serum, fixed tissue samples, frozen tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Donors: Living liver donors. This label may also refer to those evaluated for liver donation who did not go on to donate, i.e., potential living liver donors.
- Recipients: Liver transplant recipients (either living or deceased donor). This label may also refer to those who were evaluated for liver transplantation, but never received a transplant, i.e., potential recipients.

SUMMARY:
There are two principal purposes of this study: 1) to determine whether it is more beneficial for a liver transplant recipient candidate to pursue a living donor liver transplant (LDLT) or wait for a deceased donor liver transplant (DDLT), and 2) to study the impact of liver donation on the donor's health and quality of life.

DETAILED DESCRIPTION:
Adult to adult living donor liver transplantation (LDLT) is a relatively new procedure increasingly used at major transplantation centers. Relatively small numbers of cases are performed at any one center and approaches to the patient and donor are too diverse across centers to provide reliable and generalizable information on donor and recipient outcomes from individual centers. Therefore, a network of nine leading liver transplantation centers and a data coordination center (DCC) has been organized to accrue and follow sufficient numbers of patients being considered for and undergoing LDLT to provide generalizable results from adequately powered studies. This network has established the Adult to Adult Living Donor Liver Transplantation Cohort Study (A2ALL) that will conduct both retrospective and prospective studies of LDLT.

The primary study objective is to analyze the effect of choosing to pursue living liver donation. The principal hypothesis is that pursuit of a living liver allograft leads to decreased pre-transplant morbidity and mortality and better long term outcomes for patients starting from the point at which listed patients have a potential donor evaluated (at least a history and physical examination). Emerging data suggest that LDLT provides an inferior graft because of reduced parenchymal mass and added technical complexity when compared to a whole liver used for DDLT. The magnitude of the disadvantage to the LDLT graft will be assessed by comparing results between LDLT and DDLT from the time of transplant. Finally, a careful and detailed series of studies of potential and actual living liver donors is included as a primary objective because of the tremendous importance of this issue to our understanding of the impact of the procedure.

Secondary objectives will address selected biological and clinical issues in transplantation structured around the comparison between DDLT and LDLT.

ELIGIBILITY:
Inclusion Criteria - Potential Recipients:

* Potential recipient listed for single organ (liver) transplantation
* Patient is eligible for LDLT
* Age ≥ 18 years old at the time of donor history and physical exam
* Indication for transplant: non-fulminant liver disease
* Potential donor scheduled for evaluation (history and physical examination) within four weeks

Inclusion Criteria - Potential Donors:

* Meet donor criteria of the transplant center
* Age >= 18 years old at donation
* Be evaluated with a history and physical examination at the transplant center
* Potential donor's recipient listed for single organ (liver) transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential recipients and donors for transplantation will be evaluated and invited to participate in the study if they are eligible for LDLT using standard criteria for this procedure according to the practice of the transplant center.
Sampling Method: Non-Probability Sample
Enrollment: 2470 (Actual)
Dates: Start 2004-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Survival of the potential liver transplant recipient | Time from living donor evaluation to death
  Time from evaluation of a living liver donor until death of the potential recipient, to test the benefit of living liver donation.

SECONDARY OUTCOMES:
Recipient survival from time of transplant (either living or deceased donor) | From transplant until death or last follow-up
  Recipient survival from transplant to death. The goal is to compare survival among living donor versus deceased donor recipients.

OTHER OUTCOMES:
Donor complications | From the time of donation until last follow-up
  Donor complications are recorded, and graded using the Clavien scale.
Recipient complications | From time of transplantation until last follow-up
  Recipient complications are recorded, and graded using the Clavien scale.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Merion, MD, Study Chair — University of Michigan - A2ALL Data Coordinating Center; Carl L Berg, MD, Study Chair — University of Virginia Health System; Jean Emond, MD, Study Chair — Columbia University
Locations (9):
- United States (9):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Health System, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Result] Berg CL, Abecassis M, Brown RS, Everhart JE, Gillespie BW, Hulbert-Shearon TE, Merion RM. Living donor liver transplantation reduces the risk of death of transplant candidates. Hepatology 2004; 40(4)(Suppl 1): 209A.
- [Result] Ghobrial RM, Freise CE, Trotter JF, Tong L, Ojo AO, Fair JH, Fisher RA, Emond JC, Koffron AJ, Pruett TL, Olthoff KM; A2ALL Study Group. Donor morbidity after living donation for liver transplantation. Gastroenterology. 2008 Aug;135(2):468-76. doi: 10.1053/j.gastro.2008.04.018. Epub 2008 Apr 22. PMID 18505689
- [Result] Berg CL, Gillespie BW, Merion RM, Brown RS Jr, Abecassis MM, Trotter JF, Fisher RA, Freise CE, Ghobrial RM, Shaked A, Fair JH, Everhart JE; A2ALL Study Group. Improvement in survival associated with adult-to-adult living donor liver transplantation. Gastroenterology. 2007 Dec;133(6):1806-13. doi: 10.1053/j.gastro.2007.09.004. Epub 2007 Sep 14. PMID 18054553
- [Result] Freise CE, Gillespie BW, Koffron AJ, Lok AS, Pruett TL, Emond JC, Fair JH, Fisher RA, Olthoff KM, Trotter JF, Ghobrial RM, Everhart JE; A2ALL Study Group. Recipient morbidity after living and deceased donor liver transplantation: findings from the A2ALL Retrospective Cohort Study. Am J Transplant. 2008 Dec;8(12):2569-79. doi: 10.1111/j.1600-6143.2008.02440.x. Epub 2008 Oct 24. PMID 18976306
- [Result] Abecassis MM, Fisher RA, Olthoff KM, Freise CE, Rodrigo DR, Samstein B, Kam I, Merion RM; A2ALL Study Group. Complications of living donor hepatic lobectomy--a comprehensive report. Am J Transplant. 2012 May;12(5):1208-17. doi: 10.1111/j.1600-6143.2011.03972.x. Epub 2012 Feb 15. PMID 22335782
- [Result] Berg CL, Merion RM, Shearon TH, Olthoff KM, Brown RS Jr, Baker TB, Everson GT, Hong JC, Terrault N, Hayashi PH, Fisher RA, Everhart JE. Liver transplant recipient survival benefit with living donation in the model for endstage liver disease allocation era. Hepatology. 2011 Oct;54(4):1313-21. doi: 10.1002/hep.24494. PMID 21688284
- [Result] Campsen J, Blei AT, Emond JC, Everhart JE, Freise CE, Lok AS, Saab S, Wisniewski KA, Trotter JF; Adult-to-Adult Living Donor Liver Transplantation Cohort Study Group. Outcomes of living donor liver transplantation for acute liver failure: the adult-to-adult living donor liver transplantation cohort study. Liver Transpl. 2008 Sep;14(9):1273-80. doi: 10.1002/lt.21500. PMID 18756453
- [Result] Everson GT, Terrault NA, Lok AS, Rodrigo del R, Brown RS Jr, Saab S, Shiffman ML, Al-Osaimi AM, Kulik LM, Gillespie BW, Everhart JE; Adult-to-Adult Living Donor Liver Transplantation Cohort Study. A randomized controlled trial of pretransplant antiviral therapy to prevent recurrence of hepatitis C after liver transplantation. Hepatology. 2013 May;57(5):1752-62. doi: 10.1002/hep.25976. Epub 2013 Jan 17. PMID 22821361
- [Result] Fisher RA, Kulik LM, Freise CE, Lok AS, Shearon TH, Brown RS Jr, Ghobrial RM, Fair JH, Olthoff KM, Kam I, Berg CL; A2ALL Study Group. Hepatocellular carcinoma recurrence and death following living and deceased donor liver transplantation. Am J Transplant. 2007 Jun;7(6):1601-8. doi: 10.1111/j.1600-6143.2007.01802.x. PMID 17511683
- [Result] Gillespie BW, Merion RM, Ortiz-Rios E, Tong L, Shaked A, Brown RS, Ojo AO, Hayashi PH, Berg CL, Abecassis MM, Ashworth AS, Friese CE, Hong JC, Trotter JF, Everhart JE; A2ALL Study Group. Database comparison of the adult-to-adult living donor liver transplantation cohort study (A2ALL) and the SRTR U.S. Transplant Registry. Am J Transplant. 2010 Jul;10(7):1621-33. doi: 10.1111/j.1600-6143.2010.03039.x. Epub 2010 Feb 25. PMID 20199501
- [Result] Kulik LM, Fisher RA, Rodrigo DR, Brown RS Jr, Freise CE, Shaked A, Everhart JE, Everson GT, Hong JC, Hayashi PH, Berg CL, Lok AS; A2ALL Study Group. Outcomes of living and deceased donor liver transplant recipients with hepatocellular carcinoma: results of the A2ALL cohort. Am J Transplant. 2012 Nov;12(11):2997-3007. doi: 10.1111/j.1600-6143.2012.04272.x. Epub 2012 Sep 20. PMID 22994906
- [Result] Merion RM, Shearon TH, Berg CL, Everhart JE, Abecassis MM, Shaked A, Fisher RA, Trotter JF, Brown RS Jr, Terrault NA, Hayashi PH, Hong JC; A2ALL Study Group. Hospitalization rates before and after adult-to-adult living donor or deceased donor liver transplantation. Ann Surg. 2010 Mar;251(3):542-9. doi: 10.1097/SLA.0b013e3181ccb370. PMID 20130466
- [Result] Northup PG, Abecassis MM, Englesbe MJ, Emond JC, Lee VD, Stukenborg GJ, Tong L, Berg CL; Adult-to-Adult Living Donor Liver Transplantation Cohort Study Group. Addition of adult-to-adult living donation to liver transplant programs improves survival but at an increased cost. Liver Transpl. 2009 Feb;15(2):148-62. doi: 10.1002/lt.21671. PMID 19177435
- [Result] Olthoff KM, Merion RM, Ghobrial RM, Abecassis MM, Fair JH, Fisher RA, Freise CE, Kam I, Pruett TL, Everhart JE, Hulbert-Shearon TE, Gillespie BW, Emond JC; A2ALL Study Group. Outcomes of 385 adult-to-adult living donor liver transplant recipients: a report from the A2ALL Consortium. Ann Surg. 2005 Sep;242(3):314-23, discussion 323-5. doi: 10.1097/01.sla.0000179646.37145.ef. PMID 16135918
- [Result] Olthoff KM, Abecassis MM, Emond JC, Kam I, Merion RM, Gillespie BW, Tong L; Adult-to-Adult Living Donor Liver Transplantation Cohort Study Group. Outcomes of adult living donor liver transplantation: comparison of the Adult-to-adult Living Donor Liver Transplantation Cohort Study and the national experience. Liver Transpl. 2011 Jul;17(7):789-97. doi: 10.1002/lt.22288. PMID 21360649
- [Result] Shaked A, Ghobrial RM, Merion RM, Shearon TH, Emond JC, Fair JH, Fisher RA, Kulik LM, Pruett TL, Terrault NA; A2ALL Study Group. Incidence and severity of acute cellular rejection in recipients undergoing adult living donor or deceased donor liver transplantation. Am J Transplant. 2009 Feb;9(2):301-8. doi: 10.1111/j.1600-6143.2008.02487.x. Epub 2008 Dec 15. PMID 19120082
- [Result] Terrault NA, Shiffman ML, Lok AS, Saab S, Tong L, Brown RS Jr, Everson GT, Reddy KR, Fair JH, Kulik LM, Pruett TL, Seeff LB; A2ALL Study Group. Outcomes in hepatitis C virus-infected recipients of living donor vs. deceased donor liver transplantation. Liver Transpl. 2007 Jan;13(1):122-9. doi: 10.1002/lt.20995. PMID 17192908
- [Result] Trotter JF, Hill-Callahan MM, Gillespie BW, Nielsen CA, Saab S, Shrestha R, Talamantes MM, Weinrieb RM; A2ALL Study Group. Severe psychiatric problems in right hepatic lobe donors for living donor liver transplantation. Transplantation. 2007 Jun 15;83(11):1506-8. doi: 10.1097/01.tp.0000263343.21714.3b. PMID 17565325
- [Result] Trotter JF, Wisniewski KA, Terrault NA, Everhart JE, Kinkhabwala M, Weinrieb RM, Fair JH, Fisher RA, Koffron AJ, Saab S, Merion RM; A2ALL Study Group. Outcomes of donor evaluation in adult-to-adult living donor liver transplantation. Hepatology. 2007 Nov;46(5):1476-84. doi: 10.1002/hep.21845. PMID 17668879
- [Result] Trotter JF, Gillespie BW, Terrault NA, Abecassis MM, Merion RM, Brown RS Jr, Olthoff KM, Hayashi PH, Berg CL, Fisher RA, Everhart JE; Adult-to-Adult Living Donor Liver Transplantation Cohort Study Group. Laboratory test results after living liver donation in the adult-to-adult living donor liver transplantation cohort study. Liver Transpl. 2011 Apr;17(4):409-17. doi: 10.1002/lt.22246. PMID 21445924
- [Derived] Olthoff KM, Smith AR, Abecassis M, Baker T, Emond JC, Berg CL, Beil CA, Burton JR Jr, Fisher RA, Freise CE, Gillespie BW, Grant DR, Humar A, Kam I, Merion RM, Pomfret EA, Samstein B, Shaked A. Defining long-term outcomes with living donor liver transplantation in North America. Ann Surg. 2015 Sep;262(3):465-75; discussion 473-5. doi: 10.1097/SLA.0000000000001383. PMID 26258315
- [Derived] Wolf JH, Holmes MV, Fouraschen S, Keating BJ, Baker T, Emond J, Rader DJ, Shaked A, Olthoff KM. Serum lipid expression correlates with function and regeneration following living donor liver transplantation. Liver Transpl. 2016 Jan;22(1):103-10. doi: 10.1002/lt.24220. PMID 26202132
- [Derived] Everson GT, Hoefs JC, Niemann CU, Olthoff KM, Dupuis R, Lauriski S, Herman A, Milne N, Gillespie BW, Goodrich NP, Everhart JE. Functional elements associated with hepatic regeneration in living donors after right hepatic lobectomy. Liver Transpl. 2013 Mar;19(3):292-304. doi: 10.1002/lt.23592. PMID 23239552